CLINICAL TRIAL: NCT02985892
Title: Effects of Association of Trunk Stretching and Segmental Stabilization Exercises in Chronic Unspecific Low Back Pain: a Randomized Clinical Trial
Brief Title: Effects of Association of Trunk Stretching and Segmental Stabilization Exercises in Chronic Unspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Federal University of Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EATSSSE
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain
Keywords: Physical therapy; Muscle Stretching Exercises; Low Back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SSASG (Experimental): Stabilization and stretching group, 12 session, 60 minutes each. This group will perform stretching for back muscles in different positions, associated with stabilization exercises using a protocol developed by Richardson, 2005.
  Interventions: Other: SSASG
- SSPSG (Experimental): Stabilization Group, 12 session, 60 minutes each. This group will perform placebo stretching for upper limb muscles (the muscle is not stretched in it maximum extent) with stabilization exercises, using a protocol developed by Richardson, 2005.
  Interventions: Other: SSPSG

INTERVENTIONS:
Other: SSASG — Both groups will perform segmental stabilization exercises (SS), which emphasis is for the lumbar multifidus muscles (ML) and transversus abdominis (TAR), using protocol proposed by Richardson et al. Four types of exercises will be carried out with four sets of ten exercises. Muscle contractions will be held for ten seconds and followed by ten seconds rest. Between each type of exercise patients will rest for one-minute interval.
  Patients of segmental stabilization active stretching group (SSASG) will perform stretch exercises in four sets of 30 seconds for each muscle. The active stretching exercises will last 15 minutes. The muscles that will be stretched are pectorals, latissimus dorsi, latissimus dorsi, teres major, rectus abdominis, external and internal oblique.
  Arms: SSASG
Other: SSPSG — Both groups will perform segmental stabilization exercises (SS), which emphasis is for the lumbar multifidus muscles (ML) and transversus abdominis (TAR), using protocol proposed by Richardson et al. Four types of exercises will be carried out with four sets of ten exercises. Muscle contractions will be held for ten seconds and followed by ten seconds rest. Between each type of exercise patients will rest for one-minute interval.
  Patients of segmental stabilization placebo stretching group (SSPSG) will perform exercises that simulate stretching, but the muscles will not suffer effective stretch. The placebo stretching exercises will last 15 minutes. The muscles that will be stretched are wrist flexors and extensors muscles and fingers flexors and extensors muscles.
  Arms: SSPSG

SUMMARY:
The incidence of chronic nonspecific low back pain is the highest in the world population and can lead to disability. One of the standards treatments for this condition is the segmental stabilization exercises, as well as trunk stretching. However, there is no study that associates these two treatments for nonspecific low back pain. This study will be a controlled clinical trial, randomized, prospective, single-blind with a quantitative approach that compares the efficacy of the association between segmental stabilization + trunk stretching with segmental stabilization + placebo stretching in patients with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
BACKGROUND: Chronic nonspecific low back pain (LCI) has a high incidence in the world population and can lead to disability. Several therapeutic approaches have been studied to treat this pathology, but most investigate only the efficacy of one form of treatment per group. Studies show the effect of Segmental Stabilization in patients with LCI, but there is a gap on the effects of the association of trunk stretches with segmental stabilization exercises on pain and disability with LCI. Therefore, the objective of this study is to investigate the effects of the association of trunk stretching and segmental stabilization exercises on chronic non-specific low back pain in the short and medium term.

Method / Design: It will be a controlled, randomized, prospective, blinded clinical trial with quantitative approach, performed at the Clinical School of Physiotherapy of the UFPB. Participants in the study were 34 subjects of both sexes, aged 18 to 80 years, with pain equal to or greater than 3 by the Numerical Pain Scale (0/10) randomized into two groups: Placebo Stretching Group + Segmental Stabilization (n = 17) who will only do exercises of placebo stretching and segmental stabilization; And Segmental Stretching-Stabilization Group (n = 17), submitted to segmental stabilization exercises associated with trunk stretches; Both groups with 12 sessions. The results on pain intensity, functional capacity, overall effect perception, and clinical-psycho-functional assessment, as per the IMMPACT recommendations for clinical trials of effectiveness and efficacy of treatment for chronic pain, will be made by a blind After the intervention, three and six months after randomization.

Discussion: Because of its design, it will be possible to blind the evaluator, the randomizer, and the patient. At the end of the research we hope to contribute to the clinical decision-making process in the choice of therapies that improve pain and disability in patients with non-specific chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with nonspecific chronic low back pain without radicular symptoms for a period exceeding 12 months,
* pain intensity greater than 3/10 points in Numerical Pain Scale

Exclusion Criteria:

* patients who have some contraindication to perform exercises according to the American College of Sports Medicine guidelines, such as severe spinal disease (nonunion or malunion, tumors and inflammatory diseases);
* spine surgeries;
* degenerative or inflammatory disorders of the shoulder;
* patients who are in labor dispute; or are doing other types of physical therapy or drug treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in pain through Pain visual analogue scale | Before the treatment and after the treatment (immediately after the treatment, and 3 and 6 months after treatment)

SECONDARY OUTCOMES:
Global Perceived Effect Scale | Before the treatment and after the treatment (immediately after the treatment, and 3 and 6 months after treatment)

OTHER OUTCOMES:
Beck Depression Inventory | Before the treatment and after the treatment (immediately after the treatment, and 3 and 6 months after treatment)
Visual analogue scale for anxiety | Before the treatment and after the treatment (immediately after the treatment, and 3 and 6 months after treatment)
Symptoms and Adverse events or side effects | Before the treatment and after the treatment (immediately after the treatment, and 3 and 6 months after treatment)
Instrument for Measuring Patient Satisfaction (MedRisk) | Before the treatment and after the treatment (immediately after the treatment, and 3 and 6 months after treatment)
Roland Morris Disability Questionnaire | Before the treatment and after the treatment (immediately after the treatment, and 3 and 6 months after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Casarotto, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Carina Carvalho Correia Coutinho, João Pessoa, Paraíba
  - Carina Carvalho, João Pessoa, Paraíba

IPD SHARING:
Plan to Share IPD: No